CLINICAL TRIAL: NCT02224170
Title: Comparison of Effect on Quality of Recovery Outcome Between Systemic Lidocaine and Dexamethasone in Patients Undergoing Laparoscopic Cholecystectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulties in recruiting the subjects.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2014-0530
Record Dates: First submitted 2014-08-19; First posted 2014-08-25 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Gallbladder Polyp; Asymptomatic Gallstones Without Cholecystitis
Keywords: Dexamethasone; Lidocaine; Quality of Recovery; Laparoscopic cholecystectomy
MeSH Terms: interventions — Lidocaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine group (Experimental)
  Interventions: Drug: Lidocaine
- Dexamethasone group (Active Comparator)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Lidocaine — Lidocaine 2mg Kg-1 in normal saline (total volume 25mL) was infused after tracheal intubation, and lidocaine was infused at the rate of lidocaine 2mg Kg-1 h-1 (0.2 ml Kg-1 h-1, equivalent volume as normal saline in dexamethasone group) until the end of surgery (at the time of skin closure).
  Arms: Lidocaine group
Drug: Dexamethasone — Dexamethasone 8mg in normal saline (total volume 25mL) was infused after tracheal intubation, and normal saline was continuously infused at the rate of 0.2 ml Kg-1 h-1 until the end of surgery (at the time of skin closure).
  Arms: Dexamethasone group

SUMMARY:
The primary purpose of this study is to compare the effect of lidocaine and dexamethasone on postoperative quality of recovery after laparoscopic cholecystectomy

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients aged between 20 and 65 year undergoing laparoscopic cholecystectomy due to gallbladder polyp or asymptomatic gallstones without cholecystitis

Exclusion Criteria:

1. Steroid therapy or immunocompromised patients
2. Diabetes mellitus
3. Allergy to lidocaine or dexamethasone
4. Severe renal dysfunction (serum creatinine more than 1.6mg/dl)
5. Severe liver disease ( liver enzymes more than two times normal values)
6. History of atrioventricular block
7. Have a difficulty in understanding QoR-40 (40-item quality-of-recovery scoring system) or Korean language
8. History of physicologic disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
QoR-40 score | from baseline to 3 hours on the day after surgery
  40-item quality-of-recovery scoring system

SECONDARY OUTCOMES:
Incidence and severity of postoperative nausea and vomiting | from baseline to 3 hours on the day after surgery
  10 cm-visual analogue scale

OTHER OUTCOMES:
Time to first analgesic request | from baseline to 3 hours on the day after surgery
Number of rescue pain reliever | from baseline to 3 hours on the day after surgery
Severity of postoperative pain | from baseline to 3 hours on the day after surgery
  10 cm-visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Seoul, Korea, Seoul, South Korea